CLINICAL TRIAL: NCT01840241
Title: Effect of Sodium Bicarbonate on Prevention of Acute Kidney Injury in High Risk Patients Undergoing Off-pump Coronary Artery Bypass (OPCAB)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 4-2012-0419
Record Dates: First submitted 2013-04-17; First posted 2013-04-25 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Acute Kidney Injury
Keywords: sodium bicarbonate; acute kidney injury; OPCAB
MeSH Terms: conditions — Acute Kidney Injury | interventions — Sodium Bicarbonate; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BIVON group (Experimental)
  Interventions: Drug: sodium bicarbonate
- Placebo group (Placebo Comparator): normal saline infusion
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: sodium bicarbonate — BIVON group were received 0.5 mmol/kg of sodium bicarbonate for 1hours after induction of anesthesia and following 0.15 mmol/kg of sodium bicarbonate during the operation.
  Arms: BIVON group
Drug: normal saline
  Arms: Placebo group

SUMMARY:
In this single-site, randomized, controlled and double-blind clinical trial, the investigators evaluate the effect of sodium bicarbonate on prevention of acute kidney injury in high risk patients undergoing off pump coronary bypass surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 20 years
* scheduled for elective coronary artery bypass grafting.
* preoperative estimated glomerular filtration rate (eGFR) : 30 ~ 89 %
* LVEF < 35%
* NYHA class III or IV
* age > 70
* DM
* reoperation

Exclusion Criteria:

* acute renal impairment
* patients who receive dialysis
* patients who receive steroid ( > 10mg/day prednisolon or equivalent)
* hemo-alkalosis
* hypernatremia
* pulmonary edema
* Hemoglobin < 10 mg/dL

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2015-10-20 (Actual); Study Completion 2015-10-20 (Actual)

PRIMARY OUTCOMES:
compare the incidence of acute kidney injury | Change of Indexes of renal function including SCr, cystatin C, creatinine clearance from 24 hrs before operation to postoperative day (POD) 5.
  The diagnostic criteria for AKI is followed by AKIN criteria (absolutely increase in the SCr concentration ≥ 0.3 mg/dL from baseline, ≥ 50% increase in the SCr concentration within 48 hours after operation).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of anesthesiology and pain medicine, Seoul, South Korea

REFERENCES:
- [Derived] Soh S, Song JW, Shim JK, Kim JH, Kwak YL. Sodium bicarbonate does not prevent postoperative acute kidney injury after off-pump coronary revascularization: a double-blinded randomized controlled trial. Br J Anaesth. 2016 Oct;117(4):450-457. doi: 10.1093/bja/aew256. Epub 2016 Oct 17. PMID 28077531